CLINICAL TRIAL: NCT06618326
Title: ACUPUNCTURE VERSUS BIOFEEDBACK TRAINING ON BOWEL MOTILITY IN CHILDREN WITH FUNCTIONAL CONSTIPATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, ahmed fekry salman, Al-Ahliyya Amman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: acupuncture versus biofeedback
Record Dates: First submitted 2024-09-17; First posted 2024-10-01 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-02

CONDITIONS: Constipation - Functional
Keywords: CONSTIPATION; BIOFEEDBACK; ACUPUNCTURE
MeSH Terms: conditions — Constipation | interventions — Acupuncture Therapy; Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupuncture (Experimental): Group (A): will receive acupuncture in addition to non-pharmacological treatment advice from health care authorities such as the British Nutrition Foundation includes increasing fluid intake, physical activity and increasing dietary fiber consumption to a recommended daily intake of 30 g.
  Interventions: Device: Acupuncture
- biofeedback training (Experimental): Group (B): will receive biofeedback training in addition to non-pharmacological treatment advice from health care authorities such as the British Nutrition Foundation includes increasing fluid intake, physical activity and increasing dietary fiber consumption to a recommended daily intake of 30 g.
  Interventions: Device: biofeedback

INTERVENTIONS:
Device: Acupuncture — Twenty patients were suffering from functional constipation. They ranged in age from 7-15 years. All children had reasonable cognitive functions, and a reasonable IQ so as were able to follow the instructions. All received acupuncture regardless of the number of acupuncture points, frequency, and courses of treatment in addition to non-pharmacological treatment advice from health care authorities such as the British Nutrition Foundation includes increasing fluid intake, physical activity and increasing dietary fiber consumption to a recommended daily intake of 30 g
  Arms: acupuncture
Device: biofeedback — Twenty patients were suffering from functional constipation. They ranged in age from 7-15 years. All children had reasonable cognitive functions, and a reasonable IQ so as were able to follow the instructions. All received biofeedback training in addition to non-pharmacological treatment advice from health care authorities such as the British Nutrition Foundation includes increasing fluid intake, physical activity and increasing dietary
  Arms: biofeedback training

SUMMARY:
: Functional constipation is the most common gastrointestinal disorder affecting about 14 % of the global population and it negatively impacts the quality of life of those affected (Suares and Ford,2011). In addition, there is a substantial cost to health care systems and further out of pocket costs are incurred by those suffering from the condition. In the UK, costs of £168 million to the National Health Service have been reported by the Bowel Interest Group for just 1 year (2018-2019), with more than 175 000 patient days spent in hospital and numbers are increasing (Bowel Interest Group, 2020).

Traditional Chinese medicine believes that constipation is mostly caused by improper diet, emotional disorders, old age and physical weakness, and feelings of external evil; the disease is mainly in the intestine and is related to the spleen, stomach, lung, liver, kidney, and other visceral dysfunctions; the basic pathogenesis is the conduction dysfunction of the large intestine. Acupuncture and moxibustion treatment of constipation should start from the diseased part and the associated viscera, and the treatment principle is to clear the organs and lead the stagnation. The most used acupuncture points for the treatment of constipation in modern acupuncture are Tianshu (526 times), followed by Shangjuxu (366 times), Dachangshu (334 times), Zusanli (328 times), and Zhigou (306 times). Among them, Tianshu acupoint is the most used acupoint and it has a large gap with the value of Shangjuxu in the second place. The values of the acupoints in the 2nd to the 5th place are more balanced, and the value of Qihai in the sixth place is different from Zhigou in the fifth place. Also, the difference between the 6th and 15th positions is more balanced. From the frequency of acupuncture treatment of constipation, the top 5 acupoints are Tianshu, Shangjuxu, Dachangshu, Zusanli, and Zhigou (Fengzhi et al., 2023).

Biofeedback Therapy The goal of neuromuscular training using biofeedback techniques is to restore a normal pattern of defecation. Neuromuscular training or biofeedback therapy is an instrument-based learning process that is based on "operant conditioning" techniques. The governing principal is that any behaviour-be it a complex manoeuvre such as eating or a simple task such as muscle contraction-when reinforced its likelihood of being repeated and perfected increases several fold. In patients with dyssynergic defecation, the goal of neuromuscular training is two-fold. (Rao, 2008).

ELIGIBILITY:
Inclusion Criteria:

* children suffering from functional constipation using guidelines or the Rome IV/III/II criteria,
* Their ages ranged between 6 and 15 years.
* All children had reasonable cognitive functions, and a reasonable IQ so as were able to follow the instructions.

Exclusion Criteria:

* Exclusion Criteria were secondary constipation because of an underlying health issue or a side effect of medication use, medical conditions, psychiatric and/or neurological disorders that interfered with the gastrointestinal function and medications that influenced gastrointestinal function.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
constipation | after 12 session 3 session by week
  We limited the outcome measures to complete spontaneous bowel movement (CSBM), Bristol Stool Form Scale (BSFS), constipation symptoms scores (CSS), the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire, and Self-Rating Anxiety Scale (SAS) score. Before and after treatment, the result measurements were recorded (after 12 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No